CLINICAL TRIAL: NCT01866995
Title: Phase 3 Study of Phytotherapy "Raylis" In Congestive Processes Of The Pelvic Organs (Prostatostasis)Caused By Decrease Of Sexual Activity In Men.
Brief Title: Efficacy Study of Phytotherapy "Raylis" In Congestive Processes Of The Pelvic Organs (Prostatostasis)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Clinic of Men's Health and Couple Longevity, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHCL-01-15052013
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Congestive Processes Of The Pelvic Organs (Prostatostasis); Erectile Dysfunction; Sexual Function
Keywords: Ginseng; Prostatostasis; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

ARMS (3):
- Raylis (Experimental): This arm (10 men with symptoms of prostatostasis) will get "Raylis" (1 kapsule contains: ginseng root powder 50 mg, false ginseng root powder 50 mg, codonopsis root powder 50 mg, astragalus membranaceus root powder 50 mg, epimedium alpinum herbal extract 100 mg) 2 kapsules a day per 3 months
  Interventions: Drug: "Raylis"
- standard prostatostasis therapy (Active Comparator): This arm (20 men with symptoms of prostatostasis) will get the standard (pathogenetic) therapy of prostatostasis
  Interventions: Other: standard prostatostasis therapy
- Raylis plus standard prostatostasis therapy (Experimental): This arm (20 men with symptoms of prostatostasis) will get "Raylis" (1 kapsule contains: ginseng root powder 50 mg, false ginseng root powder 50 mg, codonopsis root powder 50 mg, astragalus membranaceus root powder 50 mg, epimedium alpinum herbal extract 100 mg) 2 kapsules a day per 3 months together with standard prostatostasis therapy
  Interventions: Drug: "Raylis"; Other: standard prostatostasis therapy

INTERVENTIONS:
Drug: "Raylis" — "Raylis" (1 kapsule contains: ginseng root powder 50 mg, false ginseng root powder 50 mg, codonopsis root powder 50 mg, astragalus membranaceus root powder 50 mg, epimedium alpinum herbal extract 100 mg)
  Arms: Raylis; Raylis plus standard prostatostasis therapy
Other: standard prostatostasis therapy
  Arms: Raylis plus standard prostatostasis therapy; standard prostatostasis therapy

SUMMARY:
The purpose of this study is to investigate the efficacy of Phytotherapy "Raylis" (Ginseng Root Powder 50 mg, False Ginseng Root Powder 50 mg, Codonopsis Root Powder 50 mg, Astragalus Membranaceus Root Powder 50 mg, Epimedium Alpinum Herbal Extract 100 mg) In Congestive Processes Of The Pelvic Organs (Prostatostasis) In Congestive Processes Of The Pelvic Organs (Prostatostasis)

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Symptoms of prostatostasis lasting for at least 3 months during the past 6 months:
* Pathological changes on uroflowmetry (maximum flow rate of less than 15 ml / s, average urinary flow rate of less than 12 ml / sec)
* TRUS Prostate volume more than 22 ml at TRUS
* TRUS picture of Prostatostasis
* I-PSS 7-20
* IIEF-5) - 12-21

Exclusion Criteria:

* Contraindications and limitations to use of the drug Raylis listed in the instructions for medical use *
* Diabetes mellitus (type 1 and type 2, decompensation)
* Neurogenic disorders (acute cerebral circulatory disorders, Alzheimer's disease, spinal cord injury)
* A history of pelvic trauma
* Patients who had undergone radical prostatectomy and other surgical interventions on the pelvic organs
* Concomitant use of supplements to improve the erectile function, use of the anti-androgens, anti-depressants, finasteride.
* Diagnosed BPH
* Current participation in a clinical trial and / or study medication for 30 days prior to inclusion
* Any form of substance abuse, mental disorder or condition which, in the opinion of the investigator, may complicate communication with the researcher.
* The inability or unwillingness to comply with the scheme of visits according to protocol.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
TRUS prostate | 3 months

SECONDARY OUTCOMES:
Uroflowmetry | 3 months

OTHER OUTCOMES:
IPSS | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Kalinchenko, MD PhD, Principal Investigator — Clinic of Men's Health and Couple Longevity, str Zoologicheskaya, 2-7 Moscow Russia
Locations (1):
- Clinic Of Men's Health and Couple Longevity, Moscow, Russia